CLINICAL TRIAL: NCT02730312
Title: A Phase 1 Multiple Dose Study to Evaluate the Safety and Tolerability of XmAb®14045 in Patients With CD123-Expressing Hematologic Malignancies
Brief Title: PH 1 Study to Evaluate Safety and Tolerability of XmAb14045 in Patients With CD123-expressing Hematologic Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xencor, Inc. (Industry)
Collaborators: ICON Clinical Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XmAb14045-01
Record Dates: First submitted 2016-03-31; First posted 2016-04-06 (Estimated); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: Acute Myelogenous Leukemia; B-cell Acute Lymphoblastic Leukemia; Blastic Plasmacytoid Dendritic Cell Neoplasm; Chronic Myeloid Leukemia, Blast Crisis
Keywords: AML; B-ALL; BPDCN; CML; Blast Crisis
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Burkitt Lymphoma; Blastic Plasmacytoid Dendritic Cell Neoplasm; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Blast Crisis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- XmAb14045 (Experimental): Biological/Vaccine: XmAb14045 Administered IV weekly up to 8 weeks
  Interventions: Biological: XmAb14045

INTERVENTIONS:
Biological: XmAb14045 — Administered IV weekly up to 8 weeks, with or without step-up dosing

SUMMARY:
The purpose of this study is to determine the safety and tolerability of weekly intravenous (IV) administration of XmAb14045 and to determine the maximally tolerated dose (MTD) after the first dose, and then to determine the MTD after second and subsequent infusions.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of 1 of the following diseases:

  * Primary or secondary AML (including erythroleukemia and eosinophilic leukemia, but excluding acute promyelocytic leukemia)
  * B-cell ALL
  * BPDCN
  * CML in blast phase, resistant or intolerant to tyrosine kinase inhibitor therapy
* Patients with relapsed or refractory disease with no available standard therapy
* ECOG performance status 0-2
* Not a candidate for, or refusing treatment with hematopoietic stem cell transplantation
* Fertile patients must agree to use effective contraception during and for 4 weeks after the last dose of XmAb14045
* Male patients must agree to use highly effective contraception, and refrain from donating sperm during the treatment period and for at least 4 weeks after the last dose of XmAb14045
* Able and willing to complete the entire study

Exclusion Criteria:

* Systemic antineoplastic therapy (including cytotoxic chemotherapy and toxin immunoconjugates, but excluding hydroxyurea), unconjugated antibody therapy, or radiotherapy within 2 weeks of the first dose of study treatment, or small molecule kinase inhibitors within 6 elimination half-lives of the first dose of study treatment.
* Prior therapy with CD123- or IL-3R-directed immunotherapies, including monospecific and bsAbs, immunoconjugates, or chimeric antigen receptor- modified T-cell therapy
* Failure to recover from Grade 3 or 4 toxicity from previous treatment (unrelated to malignant bone marrow involvement)
* Known uncontrolled central nervous system involvement by malignant disease
* Absolute blast count ≥10,000/mm3 or symptoms of leukostasis
* Diagnosis of promyelocytic leukemia
* Aspartate aminotransferase or alanine aminotransferase at screening >3.0 x upper limit of normal (ULN) unless considered due to leukemic organ involvement
* Bilirubin >1.5 x ULN, unless prior diagnosis and documentation of leukemic organ involvement, ongoing hemolysis, or Gilbert's syndrome
* Serum creatinine >2.0 x ULN, or estimated creatinine clearance <40mL/min
* Active heart failure or New York Heart Association Class III or IV or Objective Assessment C or D
* History or evidence of a clinically unstable/uncontrollable disorder, condition or disease other than primary malignancy, that in the opinion of the Investigator would pose a risk to the patient safety or interfere with the study evaluation, procedures, or completion
* Evidence of any active, uncontrolled bacterial, viral, parasitic, or systemic fungal infections within 1 week of first dose of study drug
* Positive test for human immunodeficiency virus (HIV) -I or -II antibodies, hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), or hepatitis C virus (HCV) antibody (unless HCV viral load test by PCR is negative). HBcAb positivity will be allowed if one or more of the following is true: a) HBsAb is present; b) hepatitis B DNA testing is negative and the patient is receiving hepatitis B reactivation prophylaxis with entecavir, tenofovir, or lamivudine
* Patient is pregnant or breast feeding, or planning to become pregnant while enrolled in the study, up to the End of Study visit
* Patients with substance abuse or other medical or psychiatric conditions that, in the opinion of the Investigator, would confound study interpretation or affect the patient's ability to tolerate or complete the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2021-09 (Actual); Study Completion 2021-09 (Actual)

PRIMARY OUTCOMES:
Safety as determined by the number of participants with treatment-related adverse events | Baseline Day 1 through Day 56
  Treatment-related adverse events as assessed by CTCAE v4.03
Identify maximum tolerated (MTD) and/or recommended dose (RD) and schedule for XmAb14045 dosing | Baseline Day 1 through Day 56
  Identify maximum tolerated (MTD) and/or recommended dose (RD) and schedule for XmAb14045 dosing

CONTACTS AND LOCATIONS:
Overall Officials: Raman Garcha, MD, Study Director — Xencor, Inc.
Locations (9):
- United States (9):
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - Blood and Marrow Transplant Group of Georgia, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - The University of Chicago Medical Center, Chicago, Illinois
  - Wexner Medical Center at The Ohio State University, Columbus, Ohio
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Swedish Cancer Institute, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ravandi F, Bashey A, Foran J, Stock W, Mawad R, Short N, Yilmaz M, Kantarjian H, Odenike O, Patel A, Garcha R, Ainsworth WB, Clynes R, Kanodia J, Ding Y, Li H, Kye S, Mims A. Phase 1 study of vibecotamab identifies an optimized dose for treatment of relapsed/refractory acute myeloid leukemia. Blood Adv. 2023 Nov 14;7(21):6492-6505. doi: 10.1182/bloodadvances.2023010956. PMID 37647601